CLINICAL TRIAL: NCT00663065
Title: An Ascending Multiple-Dose Study of the Safety, Pharmacokinetics, and Pharmacodynamics of PAZ-417 Administered Orally to Elderly Subjects
Brief Title: A Study of the Safety of PAZ-417 in Healthy Elderly Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3186A1-1102
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Healthy
Keywords: Healthy subjects over 65; healthy subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- arm 1 (Experimental)
  Interventions: Drug: PAZ-417

INTERVENTIONS:
Drug: PAZ-417

SUMMARY:
This is study to determine the safety of PAZ-417 in healthy adults over 65.

ELIGIBILITY:
Inclusion:

1. A signed and dated IRB-approved informed consent form before any study specific screening procedures are performed.
2. Ability to read English or Spanish.
3. Men or women greater than or equal to 65 years of age on study day 1. Women must be either surgically sterile (hysterectomy and/or oophorectomy) or postmenopausal for greater than or equal to 1 year (with estradiol less than or equal to 25 pg/mL[92 pmol/L] and FSH greather than or equal to 38 mIU/mL) and must have a negative serum pregnancy test result within 48 hours before administration of test article. Women who are surgically sterile must provide documentation of the procedure by an operative report or by ultrasound.
4. Subjects should have a hemoglobin level greater than or equal to 12 g/dL at the screening visit.

Exclusion

1. Any significant unstable or uncontrolled cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
2. History of vascular disorders (peripheral, coronary, venous), chronic inflammatory disorders (eg, rheumatoid arthritis), hematologic disorders, or bleeding disorders (eg, hemophilia, idiopathic thrombocytopenic purpura, VonWillebrand disease).
3. Presence or history of symptomatic vertigo, significant cardiac valvular disease, congestive heart failure, angina pectoris significant cardiac arrhythmia, or seizures.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
safety as determined by adverse events, ECGs, vitals signs, and laboratory test results | 6 months

SECONDARY OUTCOMES:
Drug distribution in the blood | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Tempe, Arizona, United States